CLINICAL TRIAL: NCT03858270
Title: Inhibition of α-synuclein Cell-cell Transmission by NMDAR Blocker, Memantine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Edwin George, MD, PhD, Associate Professor of Neurology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09282018
Record Dates: First submitted 2018-10-02; First posted 2019-02-28 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantine (Experimental): Memantine will be started at 10 mg tablet once/day for a week at bedtime. After one week Memantine will be administered at 10 mg tablet twice/day for 51 weeks.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo will be started at 10 mg tablet once/day for a week at bedtime. After one week placebo will be administered at 10 mg tablet twice/day for 51 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine will be started at 10 mg tablet once/day for a week at bedtime. After one week Memantine will be administered at 10 mg tablet twice/day for 51 weeks.
  Other Names: Namenda
  Arms: Memantine
Other: Placebo — Placebo will be started at 10 mg tablet once/day for a week at bedtime. After one week Placebo will be administered at 10 mg tablet twice/day for 51 weeks.
  Arms: Placebo

SUMMARY:
Lewy Body Dementia (LBD), is the second most common form of dementia after Alzheimer's Disease. Dementia is defined as a serious loss in cognitive ability due to damages or disease in the brain beyond what is normal aging. With Lewy Body Dementia, protein deposits, or Lewy Bodies, accumulate in nerve cells throughout the brain, affecting motor control, memory and thinking. LBD can also form with the progression of Parkinson's disease (PD). PD is a degenerative nervous system disorder that affects movement ability. Using more sensitive MRI imaging techniques the investigators are attempting to see if disease progression can be monitored more closely. At the same time, the study medication Memantine will be compared to a placebo to determine if it can be used to slow the progression of PD. The purpose of this study is to assess if disease progression can be better monitored through brain imaging and if Memantine will help slow disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with idiopathic PD for at least 2 or more years
2. 45 to 85 years of age
3. Have been on stable doses of anti-Parkinson medication
4. Able to give informed consent
5. Able to undergo brain MRI
6. Unilateral symptoms
7. A score of 26 or greater on the Montreal Cognitive Assessment (MOCA), a measure of a patients short-term memory recall, the ability to determine visual-spatial relationships of objects, attention, concentration, working memory, language and orientation to time and place
8. Use of one method of medically approved contraceptive

Exclusion Criteria:

1. History of any surgical intervention for treating PD (i.e. deep brain stimulation)
2. Extreme physical disability
3. History or current diagnosis of unstable psychiatric condition
4. Presence of dementia or any other condition that prevents the ability of the participant to provide fully informed consent
5. Other brain disease
6. Treatment with Memantine 30 days prior to baseline
7. Females who are pregnant or nursing
8. Presence of interacting medications with Memantine or co-morbid medical conditions that may be exacerbated by this agent
9. Moderately significant drug interactions with Dextromethorphan, Amantadine, Sodium Bicarbonate, and Acetazolamide
10. Previous Allergic reaction to Memantine
11. Any genetic form of PD

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Rey Auditory Verbal Learning Test (RAVLT) Scores (baseline to year-1) | Change from baseline RAVLT at year 1
  Investigate the effects of Memantine administration on the global cognitive status and executive function
Change in Trail test performance time (baseline to year-1) | Change from baseline Trail test at year 1
  Investigate the effects of Memantine administration on visual attention and task switching
Change in Stroop Color Word Test performance (baseline to year-1) | Change from baseline Stroop Color Word Test at year 1
  Investigate the effects of Memantine administration on cognitive interference and processing speed
Change Judgment of Line Orientation test performance score (baseline to year-1) | Change from baseline Judgment of Line Orientation test at year 1
  Investigate the effects of Memantine administration on visuospatial skills

SECONDARY OUTCOMES:
Change in the Intracellular volume (ICV), as measured by MRI NODDI sequence, in multiple brain regions, baseline to year-1. | Change from baseline to year-1 of ICV for each brain region mentioned above.
  ICV component is calculated from the NODDI MRI, using available software, for dorsolateral prefrontal cortex, precuneous, anterior cingulate, posterior cingulate, hippocampus, entorhinal cortex, thalamus, caudate, putamen, association visual cortex, and primary visual cortex. The change in ICV fro each region will be calculated from baseline to year-1, and would constitute a regional outcome measure, but due to the number of regions, they have all been described under outcome#5, since they have the same unit of measurement. Group comparisons (i.e. placebo v. memantine for each region) will be corrected for multiple comparisons as appropriate (E.g Bonferroni )
Change in the mean kurtosis (MK), an index of tissue complexity, as measured by MRI diffusion kurtosis (DKI) sequence sequence, in multiple brain regions (mentioned in outcome #5), baseline to year-1. | Change from baseline to year-1 of MK for each brain region mentioned above.
  MK is calculated from the DKI MRI, using available software, for regions mentioned in outcome #5. The change in MK from each region will be calculated from baseline to year-1. Group comparisons (i.e. placebo v. memantine for each region) will be corrected for multiple comparisons as appropriate (E.g Bonferroni )
Change in cortical thickness (Cth), as measured by MRI T1 sequence, in multiple brain regions (mentioned in outcome #5), baseline to year-1. | Change from baseline to year-1 of Cth for each brain region mentioned above.
  Cth is calculated from T1 MRI, using available software, for regions mentioned in outcome #5. The change in Cth from each region will be calculated from baseline to year-1. Group comparisons (i.e. placebo v. memantine, for each region) will be corrected for multiple comparisons as appropriate (E.g Bonferroni )
Change in fractional anisotropy (FA), as measured by diffusion tensor imaging (DTI) sequence, in multiple brain regions (mentioned in outcome #5), baseline to year-1. | Change from baseline to year-1 of FA for each brain region mentioned above.
  Utilizing FA to investigate white matter integrity in corpus callosum, inferior longitudinal fasciculus, and corona radiata. The change in FA from each region will be calculated from baseline to year-1. Group comparisons (i.e. placebo v. memantine, for each region) will be corrected for multiple comparisons as appropriate (E.g Bonferroni )

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States